CLINICAL TRIAL: NCT04781504
Title: Exercise Training in Women With Heart Disease: A Randomized Controlled Trial
Brief Title: Exercise Training in Women With Heart Disease
Acronym: EXCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Jennifer Reed, Principal Investigator, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20200732-01H
Record Dates: First submitted 2020-10-30; First posted 2021-03-04 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Coronary Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care + moderate-intensity continuous exercise training (Experimental): 2 days/week Warm-up: 60-70% peak HR - 10min Training: 70-85% peak HR - 35min Cool-down: 60-70% peak HR - 15min
  Interventions: Behavioral: Exercise
- standard care + high-intensity interval training (Experimental): 2 days/week Warm-up: 60-70% peak HR - 10min Training: 85-95% peak HR - 25 minutes (4x4-minutes of high-intensity intervals interspersed with 3 minutes of low-intensity intervals) Cool-down: 60-70% peak HR - 10min
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — intervention groups will complete supervised virtual exercise sessions for 12 weeks using the platform preferred by the patient (Zoom care, Zoom business, Google duo, google meet, FaceTime, join.me, WhatsApp Call, etc). The appointment will be scheduled and conducted 2 days per week. The first class will be conducted on-site to teach the patient how to take vitals and to do an in-person exercise session

SUMMARY:
Coronary heart disease (CHD) is a leading cause of premature death in Canadian women. Women who suffer an acute coronary event are more likely than men to be physically inactive, have lower exercise capacity, and die in the next year. The standard cardiac rehabilitation (CR) programs do not meet women's needs. There is a need to address these issues to increase participation in CR. The main purpose of this project is to evaluate the effects of high-intensity interval training (HIIT) compared to moderate-intensity continuous exercise training (MICE) on exercise capacity and quality of life in women with CHD. Positive results of this study will fill the gap in knowledge in exercise training, levels of motivation, self-efficacy and enjoyment following HIIT vs. MICE in women with CHD.

ELIGIBILITY:
Inclusion Criteria:

* Women with CHD (e.g. CABG or PCI at least 4 weeks but less than 12 weeks post event or procedure; acute myocardial infarction; or, stable angina with corroborating evidence of CHD);
* Patient is able to perform a symptom-limited CPET (this is needed to determine peak HR for the exercise training prescription); and,
* Patient is able to read and understand English or French.

Exclusion Criteria:

* Patient is currently participating in routine exercise training (>2x/week) (this may reduce the impact of the program on outcomes);
* Patient has: a ventricular ejection fraction <45%; unstable angina; or established diagnosis of chronic obstructive pulmonary disease, severe mitral or aortic stenosis, or hypertrophic obstructive cardiomyopathy (this may interfere with the ability to engage in MICE or HIIT);
* Patient has unmanaged psychiatric illness (e.g. active psychosis, suicidal ideation) or cognitive impairment (this may confound improvements in physical and health outcomes);
* Patient does not have internet connection;
* Patient is unable to provide written informed consent; or
* Patient is unwilling or unable to return for follow-up visits at 12 and 26 weeks.
* Patient is unwilling to be randomized to HIIT or MICE

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Change in Exercise capacity | from baseline to week-6 and from baseline to week-12
  will be measured using a gold standard symptom-limited, cardiopulmonary exercise test (CPET) on an electronically braked cycle ergometer. Gas exchange will be monitored continuously; the highest rate of oxygen uptake achieved (i.e. peak VO2 in mL/kg/min) during the last minute of the CPET will represent exercise capacity.

SECONDARY OUTCOMES:
physical and mental health | from baseline to 12 weeks and baseline to 26 weeks
  physical and mental health will be measured using the Mental Health Composite Scale (MCS) and Physical Composite Scale (PCS) of the Short Form-36 questionnaire. It consists of 36 items that contribute to eight subscales summarized into a physical component summary scale (PCS) and a mental component summary scale (MCS). A higher score on a 0-100 scale indicates a better quality of life.
Disease-specific Quality of Life, global health, physical and emotional health | from baseline to 12 weeks and baseline to 26 weeks
  measured using the HeartQoL, a validated 14-item questionnaire that assesses patients' feelings on how heart disease affects daily functioning, providing a global-health related QoL score and physical and emotional subscales. Higher score means better quality of life. Score range from 0-3, where higher scores represents better heart quality of life.
Anxiety | from baseline to 12 weeks and baseline to 26 weeks
  measured using the General Anxiety and Depression-7 (GAD-7). Score ranges from 0-21 where higher scores means a more severe level of anxiety.
Depression | from baseline to 12 weeks and baseline to 26 weeks
  measured using the Patient Health Questionnaire (PHQ-9). Scores range from 1-27 where higher scores means higher depression severity.
body composition - BMI | from baseline to 12 weeks and baseline to 26 weeks
  body mass (kg) and height (cm) will be measured to calculate body mass index (kg/m^2)
body composition - Waist circumference | from baseline to 12 weeks and baseline to 26 weeks
  Changes in body composition from baseline to 12 weeks and baseline to 26 weeks are measured by waist circumference (cm).
body composition - BIA | from baseline to 12 weeks and baseline to 26 weeks
  Changes in body composition from baseline to 12 weeks and baseline to 26 weeks are measured by bioelectrical impedance (%)
Vital Signs - Resting Blood Pressure | from baseline to 12 weeks and baseline to 26 weeks
  changes in vital signs will be measured using resting blood pressure (mmHg) in a seated position after a 5-minute rest period on the right arm using an automated monitor (BPTru) that measures 6 times (the first will be discarded and an average of the last 5 measurements will be used for statistical analyses) at 2-minute intervals.
Vital Signs - Resting Heart Rate | from baseline to 12 weeks and baseline to 26 weeks
  changes in vital signs will be measured using resting heart rate (bpm)
Self-determined motivation for exercise | from baseline to 12 weeks and baseline to 26 weeks
  the 24-item Behavioural Regulation in Exercise questionnaire (BREQ-3) yields an overall Relative Autonomy Index (RAI) score, representing overall self-determined motivation. The scale ranges from -3 "amotivation to +3 "intrinsic regulation".
Overall self-efficacy for exercise | from baseline to 12 weeks and baseline to 26 weeks
  the 9-item Multidimensional Self-Efficacy for Exercise Scale (MSES-R) yields an overall self-efficacy for exercise score reflecting scheduling, task and coping self-efficacy. The MSES consists of nine items on a 100% confidence scale ranging from 0 = "no confidence" to 100 = "completely confident."
Physical activity enjoyment | from baseline to 12 weeks and baseline to 26 weeks
  the 18-item Physical Activity Enjoyment Scale (PACES) measures the extent (on a 7-point Likert scale) to which participants enjoy doing physical activity. Overall enjoyment for physical activity score is determined by summing the items, with a range of 18-126 being possible. Higher scores indicate higher enjoyment.
Gender - TMF | from baseline to 12 weeks and baseline to 26 weeks
  using the Traditional Masculinity and Femininity scale (TMF). A score close to 4 refers to be moderately feminine and masculine.
Gender - Genesis-Praxy | from baseline to 12 weeks and baseline to 26 weeks
  using the Genesis-Praxy questionnaire.
COVID-19 Signs and Symptoms, Complications and Treatments | from baseline to 12 weeks and baseline to 26 weeks
  using a self-reported questionnaire. No score reported with this questionnaire

OTHER OUTCOMES:
Physical activity levels | from baseline to 12 weeks and baseline to 26 weeks
  will be measured objectively. The ActiGraph wGT3X-BT accelerometer (ActiGraph, Pensacola, Florida) will be worn over the right hip for 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
it is not yet known if there will be a plan to make IPD available.